CLINICAL TRIAL: NCT04502147
Title: How to Provide Vascular Control of Splenic Artery Aneurysm? Report of Two Cases
Status: Completed | Type: Observational
Sponsor: Tecnologico de Monterrey (Other)
Responsible Party: Principal Investigator, Alejandro Ruiz Velasco Santacruz, Chief of Residents, Tecnologico de Monterrey
Other Study IDs: 168/7
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Arterial Splenic Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic Splenectomy — Laparoscopic splenectomy by ligating the splenic artery

SUMMARY:
Spleen artery aneurysm represents the most common visceral aneurysm and the third most common splanchnic aneurysm. Most patients have no symptoms and are diagnosed as a part of other diagnostic focuses and examinations. The investigators present two patients with splenic artery aneurysms localized in the splenic hilum, who auspiciously undergo laparoscopic splenectomies with hem-o-lock clips in the vascular hilum without complications. These two cases showed that in addition to the numerous advantages of minimally invasive approaches, there is the possibility to improve laparoscopic technique in terms of safety and economic reasons by using hem - o - lock clips as a hemostatic technique securing the vascular elements of the splenic hilum.

ELIGIBILITY:
Inclusion Criteria:

Adults patients (>18 year old) with splenic arterial aneurysms

Exclusion Criteria:

Patients younger than 18 years old. Patients without splenic arterial aneurysms

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 41-year-old patient who was diagnosed with splenic artery enlargement on a routine ultrasound examination.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Arterial Splenic Aneurysm | July 2020
  Asses the splenic hilium after operating a splenic arterial aneurysm. It will be measure by the follow up of the patient, by consult and physical examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Tecnologico de Monterrey, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No